CLINICAL TRIAL: NCT00363376
Title: A Double-Blind, Placebo-Controlled Study of Zonisamide to Prevent Olanzapine-Associated Weight Gain
Brief Title: A Study of Zonisamide to Prevent Olanzapine-Associated Weight Gain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lindner Center of HOPE (Other)
Collaborators: Eli Lilly and Company (Industry); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 06-06-14-01; F1D-MC-X269
Record Dates: First submitted 2006-08-09; First posted 2006-08-15 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Weight Gain
Keywords: olanzapine; zonisamide; weight gain; bipolar disorder; psychotic disorders
MeSH Terms: conditions — Weight Gain; Bipolar Disorder; Psychotic Disorders | interventions — Zonisamide; Olanzapine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pill (Experimental): olanzapine and placebo ("sugar pill")
  Interventions: Drug: zonisamide; Drug: olanzapine; Drug: Sugar Pill (placebo)
- Zonisamide (Experimental): olanzapine and zonisamide (active drug)
  Interventions: Drug: zonisamide; Drug: olanzapine

INTERVENTIONS:
Drug: zonisamide — Zonisamide will be administered at an initial dose of 100 mg/d for 7 days. Subsequently, zonisamide may be increased, based on clinical response and tolerability, by 100mg/d every 7 days to a maximum of 600 mg/d by the end of the sixth week of treatment. The maximum amount of zonisamide allowed during the study will be 600 mg/day. The minimum amount of zonisamide allowed during the study will be 100 mg/d. Zonisamide will initially be given as a single pm dose, but alterations in dosing will be permitted to reduce side effects (e.g., as BID dosing to reduce nausea).
  Other Names: Zonegran
Drug: olanzapine — olanzapine will be administered open-label at 5-20 mg/d titrated to optimize response and minimize side effects
  Other Names: Zyprexa; Zydis
Drug: Zonisamide — zonisamide ranging from 100mg to 600mg daily
  Other Names: Zonegran
  Arms: Zonisamide
Drug: Sugar Pill (placebo) — sugar pill (placebo) for zonisamide
  Arms: Sugar pill

SUMMARY:
The specific aim of this study is to evaluate the efficacy, tolerability, and safety of zonisamide therapy in the prevention of weight gain associated with olanzapine treatment for psychotic or bipolar disorders.

DETAILED DESCRIPTION:
This is a single center, 16-week, randomized, double-blind, placebo-controlled, parallel group, flexible-dose study in 60 outpatients with schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, psychotic disorder NOS, or bipolar disorder types I, II, or NOS by DSM-IV-TR criteria43 with a BMI > 22 for whom treatment with olanzapine (5-20 mg/day) would be appropriate as monotherapy or adjunctive therapy. Subjects who meet entry criteria will be randomized to treatment with olanzapine plus zonisamide or olanzapine plus placebo. All subjects will receive Personal Wellness Solution Counseling (http://www.zyprexa.com/hcp/hcp_patient_c_solutions_print.jsp). Both before and after randomization to zonisamide or placebo, patients will not be permitted to have any other major psychotropic medications (antipsychotics, mood stabilizers, antidepressants, or anxiolytics) added to their medication regimens. The primary outcome measure will be change in weight. Secondary outcome measures will include the Young Mania Rating Scale (YMRS),44 the Inventory for Depressive Symptoms (IDS),45 the Positive and Negative Symptoms Scale (PANSS),46 the Clinician Global Improvement (CGI) scale,47 the Binge Eating Scale (BES) 48, BMI, waist circumference, and metabolic variables (fasting lipids, glucose, insulin).

Subjects will be inpatients or outpatients at the time of randomization to olanzapine-zonisamide or olanzapine-placebo. Throughout the study, psychiatric scales will be used to assess psychiatric symptoms, and the presence of treatment-emergent adverse events will be monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

Criteria for entering this study will include all of the following:

1. Subjects must be 18 years of age or older.
2. Subjects must have schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, psychotic disorder NOS, or bipolar I, II, or NOS disorder as defined by DSM-IV-TR criteria.
3. Subjects must have a BMI > 22.
4. Subjects must sign the Informed Consent Document after the nature of the trial has been fully explained.
5. If female, subjects must be: postmenopausal, surgically incapable of childbearing, or practicing medically acceptable effective method(s) of contraception (e.g., hormonal methods, intrauterine device) for at least one month prior to study entry and throughout the study.
6. If exposed to olanzapine in the past, subjects must be free of olanzapine for > 3 months prior to randomization to study medication.

Exclusion Criteria:

Criteria for exclusion from this study will be any of the following:

1. Subjects with clinically significant suicidal or homicidal ideation.
2. Subjects with a current DSM-IV Axis I diagnosis of delirium, dementia, amnesia, or other cognitive disorders; a psychotic or mood disorder secondary to substance use or a general medical disorder; or a DSM-IV diagnosis of a substance use disorder within the past six months.
3. Cardiovascular, endocrine, neurologic, or hematologic disease as determined by the clinical judgment of the clinical investigator. Subjects with hypo- or hyperthyroidism unless stabilized on thyroid replacement > 3 months.
4. Subjects who are allergic to or who have demonstrated hypersensitivity to or significant adverse event from olanzapine.
5. Subjects who are allergic to or who have demonstrated hypersensitivity to zonisamide.
6. Women who are pregnant or nursing.
7. Subjects who have received an experimental drug or used an experimental device within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
change in weight from baseline to endpoint | 16 weeks

SECONDARY OUTCOMES:
changes, from baseline to endpoint, in BMI | 16 weeks
changes, from baseline to endpoint, in abdominal circumference | 16 weeks
changes, from baseline to endpoint, in metabolic parameters | 16 weeks
changes, from baseline to endpoint, in clinical global improvement of psychiatric symptoms | 16 weeks
changes, from baseline to endpoint, in manic symptoms | 16 weeks
changes, from baseline to endpoint, in depressive symptoms | 16 weeks
changes, from baseline to endpoint, in psychotic symptoms | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan McElroy, MD, Principal Investigator — The Lindner Center of HOPE
Locations (1):
- The Lindner Center of HOPE, Mason, Ohio, United States

REFERENCES:
- [Result] McElroy SL, Winstanley E, Mori N, Martens B, McCoy J, Moeller D, Guerdjikova AI, Keck PE Jr. A randomized, placebo-controlled study of zonisamide to prevent olanzapine-associated weight gain. J Clin Psychopharmacol. 2012 Apr;32(2):165-72. doi: 10.1097/JCP.0b013e3182488758. PMID 22367654